CLINICAL TRIAL: NCT06738628
Title: Pilot Prospective Trial to Demonstrate Efficacy, Feasibility, and Safety of a Disposable Endoscope Platform in Third Space Endoscopic Procedures
Brief Title: Disposable Endoscope Platform in Third Space Endoscopic Procedures
Status: Not yet recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-55176
Record Dates: First submitted 2024-08-26; First posted 2024-12-17 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Achalasia; Gastroparesis
Keywords: Per-Oral Endoscopic Myotomy; Gastric Per-Oral Endoscopic Myotomy; Disposable Endoscope
MeSH Terms: conditions — Esophageal Achalasia; Gastroparesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: (Esophageal or Gastric) Per-Oral Endoscopic Myotomy — Performing Per-Oral Endoscopic Myotomy for the treatment of either achalasia of the esophagus, or gastroparesis of the stomach.
  Other Names: POEM

SUMMARY:
This is a prospective, single-arm unblinded study performed at a single tertiary center in the United States. All subjects will receive standard medical care and no experimental interventions are going to be performed. The procedures will be performed by Dr. Mohamed Othman, Dr. Salmaan Jawaid, Dr. Tara Keihanian, and Dr. Fares Ayoub. All patients undergoing third space endoscopic procedures including e-POEM and g-POEM, meeting study inclusion criteria will be screened by study coordinators for preliminary eligibility and those who meet the inclusion criteria will be approached individually for further discussion about the study and obtaining informed consent.

The goal of this prospective, pilot trial is to demonstrate the efficacy, feasibility, safety, and clinical outcomes of third space endoscopic procedures completed using a disposable endoscope platform.

DETAILED DESCRIPTION:
Over the past decade, therapeutic endoscopy has rapidly progressed giving rise to the fields of third space endoscopy and endoscopic surgery. In the foregut, esophageal per-oral endoscopic myotomy (e-POEM) has become the standard approach for achalasia with level I data supporting its use1. For gastroparesis, randomized clinical trial data 2 now supports gastric POEM (g-POEM) use for refractory cases with promising results particularly in diabetic and post-surgical patients.

Despite the remarkable advances in endoscopic therapy, there has been comparably slower progress in innovation for endoscopic platforms. In fact, current endoscope design is not significantly different from the earliest endoscopes where tip deflection is primarily controlled by rotating dials on the shaft of the endoscope and insufflation and suction are controlled by manual pressure-controlled buttons. Original fiberoptic gastroscopes were designed to facilitate diagnostic use, where the endoscopist manipulates tip-deflection dials using both hands while viewing the intestinal mucosa through a viewer, with an assistant moving the shaft of the endoscope. This same design was then adapted for colonoscopy, and later for duodenoscopy and endoscopic ultrasound. Despite significant progress in image quality, the endoscope remains a heavy device, requiring significant dexterity and musculoskeletal fitness on behalf of the endoscopist to perform endoscopy ergonomically without risking muscle injury. In addition, endoscopes require several supportive devices to function, including a separate water pump, video processor, computer screen and if needed an electrosurgical generator, making the portability of traditional endoscopic platforms quite limited.

More recently, rising concerns about infectious complications from reusable endoscopes have led to the development of several single-use endoscope platforms. A novel disposable endoscope (AMBU single-use disposable gastroscope; AMBU USA, Columbia, Md, USA) was recently approved by the U.S. Food & Drug Administration (FDA) in 2022 for use in humans. This endoscopic platform is designed for single use and comes with several advantages compared to traditional reusable endoscopes. The platform is significantly lighter, with a weight of 650 grams compared to a traditional reusable upper endoscope which weighs approximately 3900 grams. Additionally, the single use platform has a wider depth of field and significantly smaller video processor and built in portable screen. These advantages have led our group to use the endoscope for therapeutic foregut procedures including e-POEM and g-POEM with positive results. The investigators at Baylor College of Medicine most recently published a proof-of-concept experience 3 in using the disposable gastroscope for a case of e-POEM, where the significantly lighter weight of the endoscope allowed easier maneuverability and subjectively lower musculoskeletal strain for the performing endoscopist, with no negative effects on image quality or technical aspects of the procedure.

Before wider adoption, these perceived benefits need to be demonstrated in a larger, prospective trial confirming non-inferiority to historical data from reusable platforms and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years old.
2. Patients can provide informed consent.
3. Patient is referred for third space endoscopic procedure including e-POEM, g-POEM.

Exclusion Criteria:

1. Patient is < 18 years old.
2. Patient refused and/or unable to provide consent.
3. Patient is a pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years or older, not pregnant (if a woman), consenting to the study, and presents for an Esophageal POEM, or Gastric POEM will be invited to participate on this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Day 1 (procedure day)
  Defined as the ability to perform entire myotomy (procedure) with the disposable endoscope.

SECONDARY OUTCOMES:
Total Procedure Time | During Procedure
  Total recorded time to perform procedure using disposable endoscope
Intraprocedural adverse events | During Procedure
  Adverse events emerging during procedure
Satisfactory scores on Endoscopist satisfaction | Immediately following completion of the procedure
  Satisfactory survey: with endoscope maneuverability (1-5 Likert scale; 1 being "strongly disagree" to 5 being "strongly agree"), with endoscope functionality [insufflation, suction, accessory passage] (1-5 Likert scale), with endoscope image quality (1-5 Likert scale; 1 being "strongly disagree" to 5 being "strongly agree").
Scores on musculoskeletal strain survey | Immediately following completion of the procedure
  Musculoskeletal Strain survey: Focused on Overall strain, wrist strain, shoulders strain, and neck strain

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Othman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD to other researchers.